CLINICAL TRIAL: NCT03586076
Title: A Double-Blind Randomised 2-Arm, 2-Period Crossover Study to Access the Similarity of Safety and Pharmacokinetics of JHL1922 and Pulmozyme® After Single and Repeated Administration in Healthy Subjects
Brief Title: A Comparative Safety and Pharmacokinetic Study of JHL1922 and Pulmozyme® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JHL Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JHL-CLIN-1922-01
Record Dates: First submitted 2018-06-25; First posted 2018-07-13 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JHL1922 (Experimental)
  Interventions: Biological: JHL1922
- Pulmozyme (Active Comparator)
  Interventions: Biological: dornase alfa

INTERVENTIONS:
Biological: JHL1922 — Single doses of JHL1922 2.5 mg and then 10 mg per eRapid nebulizer
  Arms: JHL1922
Biological: dornase alfa — Single doses of Pulmozyme® 2.5 mg and then 10 mg per eRapid nebulizer
  Arms: Pulmozyme

SUMMARY:
This is a double-blind, randomised, 2 single-doses and then repeated-dose (5 days), 2-arm, 2-period crossover phase 1 study in 24 healthy male or female subjects. Subjects will be randomised to one of two treatment sequences in 2 treatment periods: JHL1922 (test treatment) first and then Pulmozyme (reference treatment) or Pulmozyme (reference treatment) first and then JHL1922 (test treatment).

DETAILED DESCRIPTION:
All 24 subjects will receive either JHL1922 or Pulmozyme as single doses of 2.5 mg and then 10 mg per eRapid nebulizer, followed after a washout by a 5-period of daily dosing of 10 mg of either JHL1922 or Pulmozyme per eRapid nebulizer.

The primary objective is to assess the similarity of safety and tolerability of test products, and the exploratory objective is to assess the similarity, if possible, of the systemic levels and sputum levels of dornase alfa after administration of test products.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years, inclusive
* Body Mass Index: 18.0-30.0 kg/m2, inclusive
* Weight: between 55 and 105 kg
* Condition: healthy; normal pulmonary function by spirometry

Exclusion Criteria:

- Any medical condition that presents a potential risk to the subject and/or that may compromise the objectives of the study, incl. active, or history of, pulmonary disorders incl. asthma or chronic obstructive pulmonary disease (COPD)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 21 days
  Maximum observed concentration
AUC0-t, | up to 21 days
  Area under the concentration-time curve (AUC) up to time t, where t is the last point with concentrations above the lower limit of quantitation (calculated for single-dose treatments only)
AUC0-tau | up to 21 days
  AUC over a dosing interval tau (where tau is 24 hours, calculated for the 24 hours of Day 19 only)

CONTACTS AND LOCATIONS:
Overall Officials: Sjoerd Van Marle, MD, Principal Investigator — PRA Group B.V., a PRA Health Sciences company
Locations (1):
- JHL Biotech Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided